CLINICAL TRIAL: NCT03788655
Title: Feasibility Study on Novel Metal Stents (Moving Cell Stent) for Inoperable Tumors of the Bile Duct Tract
Brief Title: Metal Stents (Moving Cell Stent) for Inoperable Tumors of the Bile Duct Tract
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Vermehren (Other)
Collaborators: Klinikum Stadt Hanau (Other)
Responsible Party: Sponsor-Investigator, Johannes Vermehren, Record Keeper, Clinical Professor, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Other Study IDs: JWGUHMED1-010
Record Dates: First submitted 2018-12-25; First posted 2018-12-27 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Bile Duct Stricture; Bile Duct Cancer
Keywords: metal stent; biliary stricture; stenting
MeSH Terms: conditions — Bile Duct Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this feasibility study (non-randomized), the applicability of a new "moving cell" biliary stents (by HILZO) in Klatskin tumors (bile duct obstruction) will be investigated.

The HILZO Moving-Cell Stent to be examined here is a non-coated metal stent with a novelty. The meshes have a diameter of 4 mm, which is rather small compared to most other stents. This significantly increases the radial force and thus the stability of the stent. Furthermore, ingrowth by tumors in the stent is difficult. The special feature is that the individual meshes can easily be stretched to 10 mm without changing the stability of the stent. This allows a second stent to pass through the first to another segment of liver.

DETAILED DESCRIPTION:
ERCP (endoscopic retrograde cholangiopancreatography) is the standard method of treating diseases in the biliopancreatic system and the treatment goal is achieved in a very high proportion of the studies. The ERCP is based on the indirect imaging of the bile ducts by injection of contrast medium, which is visualized in X-ray fluoroscopy. Furthermore, the probing of the bile ducts by means of wire and direct interventions within the bile duct system is possible.

Malignant biliary strictures are caused by various, usually cholangiocellular or pancreatic tumors, whose surgical therapy is complex and often impossible due to advanced disease. Tumors of the papillae, lymphomas and lymph node metastases can also lead to stenosis of the extra hepatic bile ducts.

The outcome of patients with malignant biliary strictures is poor, most are already presenting with advanced disease because early symptoms are rare. In particular, the above-mentioned cholangiocellular carcinomas and pancreatic carcinomas are often resectable only in its early form with high recurrence rates. Furthermore, then only palliative concepts are possible. Various studies have shown that stenting of the biliary tract with drainage of more than 50% of the liver volume improves survival. Metal stents seem to be superior to plastic stents at a slightly higher cholangitis rate. It is therefore considered standard therapy to palliatively treat these patients with more than 3 months of life expectancy using a metal stent.

Two types of stents are currently in use, plastic stents and self-expanding metal stents (SEMS). These in turn are coated (cSEMS) and uncoated (uSEMS). In distal malignant stenosis, both cSEMS and uSEMS can be used, with a higher patency rate for cSEMS and a longer duration of uSEMS retention. The disadvantage of the uSEMS is the tumor ingrowth in the stents and the possibility of re-stenosis. Various studies have shown that metal stents are associated with better bile duct drainage and better retention time compared to plastic stents and have fewer early complications, however, a consensus regarding a survival advantage with metal stents has not yet been substantiated, with the data showing a positive trend. Since metal stents, unlike plastic stents, do not need to be changed, a significant advantage for the patient is the significant reduction in endoscopic examinations and associated hospitalization and complication rates.

The HILZO Moving-Cell Stent to be examined here is a non-coated metal stent with a novelty. The meshes have a diameter of 4 mm, which is rather small compared to most other stents. This significantly increases the radial force and thus the stability of the stent. Furthermore, ingrowth by tumors in the stent is difficult. The special feature is that the individual meshes can easily be stretched to 10 mm without changing the stability of the stent. This allows a second stent to pass through the first to another segment of liver. Previous metal stents could previously only be placed side by side in the common bile duct, thereby limiting the number of stents as a function of the gait and the stents can develop worse in the main course.

ELIGIBILITY:
Inclusion Criteria:

• Indication for the palliative metal-stent system for malignant stenosis due to biliary cancer (Klatskin tumor).

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Contraindication to an endoscopic examination
* Life expectancy under 3 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the indication for palliative stenting of the bile duct system due to non-operable Klatskin tumors type II-IV
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-12-31 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Technical feasibility of intrahepatic stenting | 12 month
  Successful biliary drainage by new stent

SECONDARY OUTCOMES:
Number of drained segments | 12
  Number of successful drained liver segments
Length of intervention | 12 month
  Length of the endoscopy with the new stent
Stent dysfunction | 12 month
  Stent migration or stenosis
Number of necessary endoscopies per year | 12 month
  Number of necessary endoscopies per year to have successful drainage
Survival rate | 12 month
  Survival of patients 12 month after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mireen Friedrich-Rust, Prof., Principal Investigator — University Clinic Frankfurt am Main
Locations (1):
- Klinikum der J. W. Goethe-Universität, Frankfurt am Main, Germany